CLINICAL TRIAL: NCT06247540
Title: Venetoclax, Rituximab and Nivolumab Combination in Patients With Richter's Transformation (RT) Arising From Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL): A Phase II Study With Safety Run-In
Brief Title: Venetoclax, Rituximab and Nivolumab in Combination for the Treatment of Richter's Transformation Arising From Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 23H01; NCI-2023-08755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00219856; NU 23H01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-12-08; First posted 2024-02-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Chronic Lymphocytic Leukemia; Richter Syndrome; Transformed Chronic Lymphocytic Leukemia to Diffuse Large B-Cell Lymphoma; Transformed Small Lymphocytic Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Nivolumab; Rituximab; CT-P10; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (venetoclax, rituximab, nivolumab) (Experimental): Patients receive venetoclax PO QD on days 1-28, nivolumab IV over 30 minutes on days 2 and 15 of cycles 1-4 and day 1 of each subsequent cycle, and rituximab IV on day 2 of cycle 1 and day 1 of cycles 2-6. Treatment repeats every 28 days up to 6 cycles in the absence of disease progression or unacceptable toxicity. After the completion of 6 cycles, rituximab is discontinued and patients receive venetoclax PO QD on days 1-28 and nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 2 years total therapy in the absence of disease progression or unacceptable toxicity. Patients undergo tissue biopsy during screening. Patients undergo a bone marrow biopsy and blood sample collection as well as PET/CT and CT or MRI during screening and on the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT, CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Nivolumab — Receive IV
  Other Names: ABP 206; BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Rituximab — Receive IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Drug: Venetoclax — Receive PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well venetoclax, rituximab and nivolumab works in treating patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) with Richter's transformation. Richter's transformation can be described as the development of an aggressive lymphoma in the setting of underlying CLL/SLL that has a very poor prognosis with conventional therapies and represents a significant unmet medical need. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Immunotherapy with monoclonal antibodies, such as rituximab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Giving venetoclax, rituximab and nivolumab together may work better than the conventional intensive immunochemotherapy to improve disease control in patients with Richter's transformation arising from CLL/SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the preliminary efficacy in terms of overall response rate (ORR) per Lugano criteria with venetoclax, nivolumab, and rituximab combination in patients with Richter's transformation.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of venetoclax, nivolumab, and rituximab combination in Richter's transformation (RT) using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).

II. To determine preliminary efficacy in terms of complete response (CR) with venetoclax, nivolumab, and rituximab combination in patients with RT.

III. To determine the preliminary efficacy in terms of minimal residual disease (MRD) negativity rate with venetoclax, nivolumab, and rituximab combination in patients with RT.

IV. To determine the preliminary efficacy in terms of progression free survival (PFS) at 12 months with venetoclax, nivolumab, and rituximab combination in patients with RT.

V. To determine the preliminary efficacy in terms of overall survival (OS) with venetoclax, nivolumab, and rituximab combination in patients with RT.

EXPLORATORY OBJECTIVES:

I. The study team will study various prognostic markers and biomarkers and correlate them with clinical response:

Ia. MRD status in bone marrow and peripheral blood; Ib. CLL prognostic markers, cytogenetics abnormalities by fluorescence in situ hybridization (FISH), IgVH mutation status, and TP53 mutation status; Ic. PD-L1 and PD-1 expression by immunohistochemistry (IHC), either in lymph node tissue samples or bone marrow; Id. T-cell subsets in the blood and tissue biopsy.

EXPLORATORY STUDIES OBJECTIVES:

I. To determine the clinical and pathological factors impacting clinical response to the rituximab-nivolumab-venetoclax combination therapy.

II. To study the role of PD-1 blockade in RT. III. To determine the role of bone marrow and peripheral blood MRD in the RT study population.

OUTLINE: This is a dose-escalation study of venetoclax.

Patients receive venetoclax orally (PO) once daily (QD) on days 1-28, nivolumab intravenously (IV) over 30 minutes on days 2 and 15 of cycles 1-4 and day 1 of each subsequent cycle, and rituximab IV on day 2 of cycle 1 and day 1 of cycles 2-6. Treatment repeats every 28 days up to 6 cycles in the absence of disease progression or unacceptable toxicity. After the completion of 6 cycles, rituximab is discontinued and patients receive venetoclax PO QD on days 1-28 and nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 2 years total therapy in the absence of disease progression or unacceptable toxicity. Patients undergo tissue biopsy during screening. Patients undergo a bone marrow biopsy and blood sample collection as well as positron emission tomography (PET)/computed tomography (CT) and CT or magnetic resonance imaging (MRI) during screening and on the trial.

After completion of study treatment, patients are followed up at 30 days and every 90 days for 5 years from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of one of Richter's transformation (to either diffuse large B cell lymphoma (DLBCL) or Hodgkin's lymphoma) with preceding CLL/SLL
* Richter's transformation refers to development of aggressive lymphoma (most commonly diffuse large B cell lymphoma (DLBCL), and less commonly Hodgkin's lymphoma) in a patient who has a pre-existing diagnosis of CLL/SLL. A pathologic diagnosis of DLBCL or Hodgkin's lymphoma in the setting of preceding CLL/SLL is required
* Patients with Richter's transformation arising from CLL/SLL may be newly diagnosed or have relapsed or progressed after prior treatment. Patients with newly diagnosed Richter transformation are eligible only if the treating physician believes they are not good candidates for standard immunochemotherapy or chemotherapy
* All patients must have measurable disease as defined by Lugano criteria 2014
* Patients must be age ≥ 18 years
* Patients must exhibit a/an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count ≥ 1,000/mcL (independent of growth factor support for ≥ 14 days) (within 14 days prior to registration)
* Platelets ≥ 30,000/mcl (independent of transfusion for ≥ 14 days) (within 14 days prior to registration)
* Hemoglobin ≥ 8 g/dL (within 14 days prior to registration)

  * Note: patients must be able to maintain this level without transfusion
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (within 14 days prior to registration)

  * Note: Autoimmune hemolytic anemia (AIHA) and Gilbert's syndrome are exceptions and bilirubin value must be < 5 x ULN
* Aspartate aminotransferase (AST) ( serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 1.5 X ULN (within 14 days prior to registration)
* Alanine transaminase (ALT) (serum glutamic-pyruvic transaminase [SPGT]) ≤ 1.5 X ULN (within 14 days prior to registration)
* Creatinine clearance ≥ 50mL/min (within 14 days prior to registration)

  * Calculate creatinine clearance (CrCl) using the Cockcroft Gault
* Patients with a known history chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a known history of hepatitis C (HCV) infection must have been treated and cure. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Females of child-bearing potential (FOCBP) must agree to adequate contraception (abstinence or acceptable methods of birth control such as barrier method or hormonal contraception) with partner(s) for the duration of study participation, for 5 months after the last dose of nivolumab and 12 months after the last dose of rituximab following completion of therapy.

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, including women who having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months; confirmation of postmenopausal state will be done by clinical history of last menstrual period)
* FOCBP must have a negative urine or serum pregnancy test within 7 days prior to registration on study.

  * NOTE: Patients are also required to have a negative pregnancy test within 24 hours of first dose of study drug
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Patients must have the ability to swallow and maintain oral medication
* Patients must be willing and able to start treatment with allopurinol or equivalent ≤ 3 days prior to starting treatment with venetoclax

Exclusion Criteria:

* Patients who have received prior nivolumab for treatment of Richter's transformation, or other PD-1/PD-L1 for the treatment of any indication.

  * Note: Prior anti-CD-20 antibody treatment is allowed with ≥ 14 day washout period. Prior treatment with nivolumab is permissible if for a different disease indication. In such cases nivolumab must have been discontinued ≥ 3 months prior to registration
* Patients who have a history of life-threatening adverse reactions attributed to compounds of similar chemical or biologic composition to venetoclax, nivolumab, or rituximab
* Patients who are refractory to venetoclax (defined by disease progression while on venetoclax or within 3 months of discontinuing venetoclax)
* Patients who have had prior chimeric antigen receptor-modified T-cell (CAR-T) therapy within the 45 days prior to registration or with any remaining CAR-T related cytokine-release syndrome or neurotoxicity
* Patients who have adverse events due to agents administered ≥ 30 days prior to registration that have not recovered to ≤ grade 2
* Patients who have had chemotherapy, radiotherapy or immunotherapy ≤ 14 days prior to registration
* Patients receiving any other investigational agents within ≤ 30 days or 5 half-lives prior to registration, whichever is shorter
* Patients who have received B-cell receptor pathway inhibitor (such as ibrutinib or idelalisib) ≤ 3 days prior to receiving study treatment
* Patients who have undergone an autologous stem cell transplant ≤ 120 days prior to registration
* Patients who have undergone an allogeneic stem cell transplant ≤ 180 days prior to registration.

  * Note: Patients must be off all immunosuppressive therapies > 30 days prior to registration, with no active graft versus host disease (GVHD)
* Patients with acute or extensive chronic graft-versus-host disease (GVHD)
* Patients who have received any of the following agents ≤ 7 days prior to receiving study treatment:

  * Steroid therapy with anti-neoplastic intent
  * Moderate or strong CYP3A inhibitors
  * Moderate or strong CYP3A inducers
* Patients who have received a live / attenuated vaccine ≤ 30 days prior to receiving study treatment
* Patients who have history of auto-immune conditions requiring ongoing or intermittent systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive medications)

  * Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients who have a history of active malignancy other than CLL/SLL or RT within the past 2 years, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri
  * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
* Patients who have known autoimmune disease or active uncontrolled autoimmune cytopenias
* Patients who have overt thyroid dysfunction (hyperthyroidism or hypothyroidism).

  * Note: Patients with chronic hypothyroidism taking stable dose of thyroid replacement therapy with normal TSH are eligible
* Patients with systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment
* Any patient who has tested positive for human immunodeficiency virus (HIV) (due to potential drug-drug interactions between anti-retroviral medications and venetoclax, as well as anticipated venetoclax mechanism based lymphopenia that may potentially increase the risk of opportunistic infections).

  * Note: HIV test is not a requirement to determine eligibility
* Patients who have malabsorption syndrome or another condition that precludes enteral route of administration
* Patients with a known contraindication or allergy to both xanthine oxidase inhibitors and rasburicase
* Patients who have a significant history of cardiovascular, pulmonary, renal, hepatic, neurologic, psychiatric, endocrinologic, metabolic, or immunologic disease that in the opinion of the investigator would adversely affect his/her participation in this study or interpretation of study results
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2029-12-29 (Estimated); Study Completion 2031-12-29 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 5 years
  Will be assessed using International Workshop on Chronic Lymphocytic Leukemia (iwCLL) and Lugano 2014 criteria for Richter's transformation (RT) patients. Will be calculated using proportions and exact 95% binomial confidence intervals.
Best response rate | Up to 5 years
  Will be assessed using iwCLL and Lugano 2014 criteria for RT patients. Will be calculated using proportions and exact 95% binomial confidence intervals.
Minimal residual disease (MRD) rate | Up to 5 years
  Will be assessed in chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) patients in the peripheral blood and bone marrow by flow cytometry, polymerase chain reaction (PCR) and/or sequencing. MRD negativity is defined as less than one CLL/SLL cell per 10,000 leukocytes (or below 10-4) on peripheral blood and/or bone marrow based flow cytometry and/or PCR based methods. Rate of MRD status will be defined as the proportion of patients who have MRD negativity status. Will be calculated using proportions and exact 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 100 days after last dose of study treatment
  Will calculate the number and percentage of toxicities by type, grade, severity and attribution. For all adverse events including laboratory values, physical examination characteristics, vital signs and electrocardiogram, Common Terminology Criteria for Adverse Events version 5.0 criteria will be used to classify the severity of the adverse event. All adverse events regardless of severity will be documented and will be summarized for regular review by the Cancer Center's Data and Safety Monitoring Committee.
Progression-free survival | Up to 5 years
  Will be assessed using iwCLL and Lugano 2014 criteria for RT patients. Will be determined using a Kaplan-Meier curves with 5-year survival and 95% confidence interval reported
Overall survival | Up to 5 years
  Will be determined using a Kaplan-Meier curves with 5-year survival and 95% confidence interval reported
Duration of response | Up to 5 years
  Will be assessed using iwCLL and Lugano 2014 criteria for RT patients. Will be summarized using median and interquartile range.
Prognostic markers and biomarkers | Up to 5 years
  Will be correlated with clinical response using a Wilcoxon rank sum test. The statistical significance of individual markers, multivariate proportional hazards regression will be used to assess multiple markers simultaneously. Prognostic markers will be related to response using Fisher's exact test or the Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Ma, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States